CLINICAL TRIAL: NCT02639143
Title: Rapid P2Y12 Receptor Inhibition Attenuates Inflammatory Cell Infiltration in Thrombus Aspirated From the Infarct-related Artery in STEMI Patients: A Prospective Randomized Trial of Ticagrelor Versus Clopidogrel
Brief Title: Rapid P2Y12 Receptor Inhibition Attenuates Inflammatory Cell Infiltration in Thrombus Aspirated From the STEMI Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-14-10167
Record Dates: First submitted 2015-11-23; First posted 2015-12-24 (Estimated); Last update posted 2021-08-23 (Actual); Status verified 2015-11

CONDITIONS: Inflammation; Thrombosis
MeSH Terms: conditions — Inflammation; Thrombosis | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ticagrelor (Experimental): Ticagrelor, 180 mg, oral administration. followed by 90 mg bid
  Interventions: Drug: ticagrelor
- Clopidogrel (Active Comparator): Clopidogrel 600 mg loading dose taken orally, followed by 75 mg qd.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: ticagrelor
  Arms: ticagrelor
Drug: Clopidogrel
  Arms: Clopidogrel

SUMMARY:
This is a prospective, randomized, parallel design study to investigate that ticagrelor could attenuate inflammatory cell infiltration in thrombus aspirated from ST elevation myocardial infarction (STEMI) patients. The anticipated duration of the study is approximately 9 months, including an anticipated enrolment period of 8 months and follow-up period of 1 month. Patients within 12 hours of symptom onset were randomly assigned in a one-to-one ratio to receive ticagrelor or clopidogrel at time of STEMI diagnosis. The primary endpoint was the extent of inflammatory cell infiltration in thrombus aspirated from STEMI patients, expressed as number of total inflammatory cells per mm2 thrombus area.

DETAILED DESCRIPTION:
This is a prospective, randomized, parallel design study to investigate that ticagrelor could attenuate inflammatory cell infiltration in thrombus aspirated from STEMI patients. The anticipated duration of the study is approximately 9 months, including an anticipated enrolment period of 8 months and follow-up period of 1 month. Patients within 12 hours of symptom onset were randomly assigned in a one-to-one ratio to receive ticagrelor or clopidogrel at time of STEMI diagnosis. The primary endpoint was the extent of inflammatory cell infiltration in thrombus aspirated from STEMI patients, expressed as number of total inflammatory cells per mm2 thrombus area.

Screening will be made to select eligible participants before intervention. Patients with documented STEMI and within 12 hours of symptom onset will be enrolled from the study site. For patients post percutaneous coronary intervention (PCI), they must be on dual-antiplatelet therapy for at least 12 months to be eligible for the study.

After the enrollment period, patients were randomly assigned in a one-to-one ratio to receive ticagrelor (180 mg loading dose) or clopidogrel (600 mg loading dose) at time of STEMI diagnosis. In addition to randomized study medication all patients should receive concomitant Ace Salicylic Acid (ASA) 100 mg daily during the treatment period according to local practice, unless they are allergic or intolerant. For those not previously given aspirin, a loading dose of 300 mg was preferred. At the end of the study, data will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Males and non-pregnant females > 18 and < 79 years of age.
* Symptoms consistent with STEMI lasting > 30 min.
* Arrival at the hospital within 12 h of the onset of chest pain.
* Intention to perform PCI

Exclusion Criteria:

* On treatment with a P2Y12 receptor antagonist (ticlopidine, clopidogrel, prasugrel, ticagrelor) in past 30 days.
* Known allergies to aspirin or ticagrelor or clopidogrel.
* On treatment with oral anticoagulant (Vitamin K antagonists, dabigatran, rivaroxaban).
* Treatment with IIb/IIIa glycoprotein inhibitors in the last 7 days.
* Known pregnancy, breast-feeding, or intend to become pregnant during the study period.
* Active pathological bleeding
* History of prior intracranial bleeding.
* Renal dysfunction (serum creatinine levels ≥ 2.0 mg/dL).
* Severe, non-catheter-related coronary artery spasm.
* New York Heart Association (NYHA) class III or IV heart failure or known left ventricular ejection fraction < 30%.
* Known severe hepatic dysfunction.
* Hemodynamic or electrical instability (including shock).
* Concomitant inflammatory diseases, malignant tumours, anaemia or thrombocytopenia.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Number of total inflammatory cells per mm2 thrombus area. | Thrombus will be got from aspiration in culprit lesions during primary PCI.It will be fixed immediately and tested in 48 hours.
  To evaluate the efficacy of ticagrelor compared to clopidogrel for the attenuation of inflammatory cell infiltration in thrombus aspirated from STEMI patients.

SECONDARY OUTCOMES:
Intracoronary thrombus size | Thrombus will be got from aspiration in culprit lesions during primary PCI.It will be fixed immediately and tested in 48 hours.
Number of neutrophils per mm2 thrombus area | Thrombus will be got from aspiration in culprit lesions during primary PCI.It will be fixed immediately and tested in 48 hours.
Number of macrophages per mm2 thrombus area | Thrombus will be got from aspiration in culprit lesions during primary PCI.It will be fixed immediately and tested in 48 hours.
Number of Myeloperoxidase-positive cells per mm2 thrombus area | Thrombus will be got from aspiration in culprit lesions during primary PCI.It will be fixed immediately and tested in 48 hours.
Serum high-sensitivity C-reactive protein level | after randomization and before loading dose P2Y12 receptor inhibitor,5-7 days after PCI,1 month ± 5 days.
  A total of three times
Plasma concentration of ticagrelor | At 90 min, 2h, 8h, 12h and 24h after received loading dose P2Y12 receptor inhibitor.
Rate of Thrombolysis In Myocardial Infarction (TIMI) major bleeding | Follow up: 1 month ± 5 days.